CLINICAL TRIAL: NCT04736524
Title: Immune Response Following COVID-19 Vaccination (IFVAC)
Brief Title: Immune Response Following COVID-19 Vaccination
Acronym: IFVAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Other Study IDs: TCAI_IFVAC
Record Dates: First submitted 2021-02-01; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: IgM and IgG in Blood
MeSH Terms: conditions — Hyper-IgM Immunodeficiency Syndrome, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rapid antibody test — Serial serology tests on day 21, 90, 180 and 365 following the first dose of the COVID-19 vaccine to detect the temporal trend of the IgM and IgG production in response to the vaccination.

SUMMARY:
Few trials have reported the safety and efficacy of the COVID-19 vaccines. However, these trials were mostly focused on post-vaccination adverse events and short-term antibody detection with none monitoring the presence of immunoglobulin G (IgG) in blood at long-term follow-up after the vaccination. This study aims to evaluate the immune response in post-vaccinated individuals across a follow-up period of one year.

DETAILED DESCRIPTION:
The COVID-19 pandemic started in December 2019 and since then has spread globally claiming over 550, 000 deaths, >12 million infections and an economic toll in the trillions of dollars to date. The urgent need for a global vaccination program to control this pandemic has prompted the development of several vaccines.

Preliminary reports from few trials evaluating the safety and efficacy of the vaccines have been published (2-4).

However, no trials have yet reported the long-term post-vaccination immune response that would potentially determine the necessity and timing for booster doses of the vaccine.

Therefore, this study is designed to assess the presence of immunoglobulin (Ig) M and G at several time points after the first and the second dose of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

• Individuals that have received first dose of COVID-19 vaccine

Exclusion Criteria:

* Unwilling to provide informed consent
* Unwilling for the follow-up serological test during the 1-year enrollment

Ages: 16 Years to 85 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individuals receiving COVID-19 vaccines
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Post-vaccination immune response | 1 year
  To assess the time for appearance and persistence of IgM and IgG after COVID-19 vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Sanghamitra Mohanty, Study Director — Texas Cardiac Arrhythmia Research Foundation
Locations (1):
- Texas Cardiac arrhythmia Institute, St. David's Hospital, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be available for research purpose only by submitting a formal request to the PI